CLINICAL TRIAL: NCT03426176
Title: The Interaction Between Oxytocin and Serotonin on the Social-emotional Brain Networks
Brief Title: The Interaction Between Oxytocin and Serotonin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-29
Record Dates: First submitted 2018-02-01; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: oxytocin; acute tryptophan depletion; emotion
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- male oxytocin and ATD group (Experimental): male subjects receiving oxytocin and ATD treatment
  Interventions: Drug: oxytocin nasal spray; Drug: ATD treatment
- male oxytocin and placebo group (Experimental): male subjects receiving oxytocin and ATD-placebo treatment
  Interventions: Drug: oxytocin nasal spray; Drug: oral placebo treatment (placebo-control for ATD)
- male placebo and ATD group (Experimental): male subjects receiving oxytocin placebo and ATD treatment
  Interventions: Drug: intranasal placebo treatment (placebo-control for oxytocin); Drug: ATD treatment
- male placebo group (Placebo Comparator): male subjects receiving oxytocin placebo and ATD placebo treatment
  Interventions: Drug: intranasal placebo treatment (placebo-control for oxytocin); Drug: oral placebo treatment (placebo-control for ATD)

INTERVENTIONS:
Drug: oxytocin nasal spray — intranasal administration of oxytocin (24 IU)
  Arms: male oxytocin and ATD group; male oxytocin and placebo group
Drug: intranasal placebo treatment (placebo-control for oxytocin) — intranasal administration of placebo nasal spray
  Arms: male placebo and ATD group; male placebo group
Drug: ATD treatment — oral administration of ATD (75.2g) (Acute Tryptophan Depletion)
  Arms: male oxytocin and ATD group; male placebo and ATD group
Drug: oral placebo treatment (placebo-control for ATD) — oral administration of a tryptophan-balanced mixture (78.2g)
  Arms: male oxytocin and placebo group; male placebo group

SUMMARY:
the study aims to explore whether there is an interaction between oxytocin and serotonin in the regulation of emotion-based behavior by using a between-subject randomized double blind pharmacological fMRI design during which 4 groups of healthy male subjects will receive combinations of oxytocin nasal-spray (versus placebo) and acute tryptophan depletion (ATD, versus placebo)

DETAILED DESCRIPTION:
Convergent evidence from animal models and human studies suggests that both, serotonin and oxytocin are important regulators of social emotional behavior. Evidence is emerging that both systems interact in this domain. To determine the interaction of both systems on human social behavior, the present study aims to combine a randomized placebo-controlled administration of modulators of both systems (Oxytocin nasal-spray and acute tryptophan depletion, ATD) and their combination within a pharmaco-fMRI experiment. To determine effects on the neural networks engaged in social emotional processing, healthy male subjects will receive single doses of oxytocin (24IU) versus placebo and ATD (75.2g) versus placebo before fMRI measures of emotion perception and resting state will be acquired. To control for potential effects of pre-medication personality traits as well as effects of medicines on mood, subjects will be administered pre-treatment assessing relevant personality traits and post-treatment assessments of mood.

ELIGIBILITY:
Inclusion Criteria:

* health subjects without past or current psychiatric or neurological disorders
* Right-handedness

Exclusion Criteria:

* History of head injury;
* Medical or psychiatric illness.
* High blood pressure, general cardio-vascular alterations
* History of drug or alcohol abuse or addiction.
* Allergy against medications or general strong allergies
* Sleep disorders.
* Visual or motor impairments

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
Neural processing during the emotion processing as assessed via fMRI | 6h after treatment
  fMRI BOLD indices of neural processing in emotion related brain regions will be compared between the treatment groups
Neural processing during the resting state as assessed via fMRI | 6h after treatment
  Resting state activity in the emotional brain networks will be compared between the treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life Science and Technology, Chengdu, Sichuan, China